CLINICAL TRIAL: NCT04085042
Title: Impact of a Multimodal Intervention on Peripheral Venous Catheterization of Cancer Patients
Acronym: MultiCat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Escola Superior de Enfermagem de Coimbra (Other)
Collaborators: Instituto Português Oncologia de Coimbra Francisco Gentil E. P. E. (Unknown)
Responsible Party: Principal Investigator, Paulo Costa, MSc, RN, Escola Superior de Enfermagem de Coimbra
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Esenfc
Record Dates: First submitted 2019-09-09; First posted 2019-09-11 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Catheterization, Peripheral
Keywords: Catheterization, Peripheral

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Usual care during peripheral venous catheterization. Nurses will continue with the normal routine practice, by preparing all needed material individually.
- PIVC pack (Experimental): Nurses will use a sterile pack that includes all needed devices for peripheral intravenous catheterization according to the latest evidence (eg, cannula, swabs, disposable tourniquet, antiseptic).
  Interventions: Device: PIVC pack

INTERVENTIONS:
Device: PIVC pack — The PIVC pack is a sterile container that includes inside all the need devices to perform peripheral catheterization. The pack is color-coded to inform healthcare professionals about the catheter caliber inside.
  Arms: PIVC pack

SUMMARY:
Peripheral intravenous catheterization (PIVC) is the most frequent invasive clinical procedure in a hospital setting, associated with significant complication rates for the patient, compromising their well-being, as well as the quality, safety, and efficacy of the care provided. The traditional approach to PIVC is considered reactive and ineffective, resulting in the exhaustion of the patients' peripheral venous access prior to consideration of other access methods and options (Moureau et al., 2012).

Evidence suggests that the safety and effectiveness of patients with a peripheral catheter are also intrinsically associated with the adequacy of materials and technologies used in clinical contexts for vein selection, as well as for catheter insertion and maintenance care (Marsh, Webster, Mihala & Rickard, 2017). Several studies point to the inadequacy of the technologies and medical devices used in this area, enhancing the occurrence of complications such as infection, phlebitis, occlusion and accidental catheter removal (Braga, 2017; Costa, 2017; Nobre & Martins, 2018).

The project investigators aim to determine whether the use of a PIVC pack will significantly reduce associated complications when compared with the usual care. Additionally, the research team aims to determine if the use of a PIVC pack will reduce the number of insertion attempts and overall procedure time, as well as improving patient and provider satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Participants who require peripheral intravenous catheterization as part of their therapeutic plan (caliber 20G or 22G);
* Participants whose primary nurse agrees to participate in the study;
* Participants who are able to give written assent or oral assent.

Exclusion Criteria:

* Confused and/or disoriented participants;
* Participants who are unable to communicate orally and/or in writing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
PIVC-related complications | This outcome will be assessed immediately following intervention, an average of 5 minutes. This outcome will be assessed through study completion, an average of 6 months
  Evaluated through a self-report scale where the nurse identifies a set of indicators associated to the occurrence of immediate complications during the procedure (extravasation, puncture of proximal anatomical structures, hematoma, etc.)

SECONDARY OUTCOMES:
Successful intravenous catheterization on the first attempt | This outcome will be assessed immediately following intervention, an average of 5 minutes. This outcome will be assessed through study completion, an average of 6 months
  Successful attempt is defined through the clear flush of the catheter with 5 mL of normal saline without extravasation.
Number of attempts to successful intravenous catheter placement | Immediately following intervention, an average of 5 minutes. This outcome will be assessed through study completion, an average of 6 months.
Time to successful placement (in minutes) | From time of randomization until the time of successful intravenous catheter placement, assessed through study completion, an average of 6 months.
Patient satisfaction | This outcome will be assessed immediately following intervention, an average of 20 minutes. This outcome will be assessed through study completion, an average of 6 months
  Evaluated through a self-report scale where the participant identifies a set of indicators associated to their satisfaction with the intervention, when compared to previous experiences.
Nurse satisfaction | This outcome will be assessed immediately following intervention, an average of 20 minutes. This outcome will be assessed through study completion, an average of 6 months
  Evaluated through a self-report scale where the nurse identifies a set of indicators associated to their satisfaction with the intervention, when compared to previous experiences.

CONTACTS AND LOCATIONS:
Overall Officials: Paulo Costa, MSc, Principal Investigator — The Health Sciences Research Unit: Nursing
Locations (1):
- Instituto Português de Oncologia de Coimbra, Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers.

REFERENCES:
- [Background] Moureau NL, Trick N, Nifong T, Perry C, Kelley C, Carrico R, Leavitt M, Gordon SM, Wallace J, Harvill M, Biggar C, Doll M, Papke L, Benton L, Phelan DA. Vessel health and preservation (Part 1): a new evidence-based approach to vascular access selection and management. J Vasc Access. 2012 Jul-Sep;13(3):351-6. doi: 10.5301/jva.5000042. PMID 22307471
- [Background] Marsh N, Webster J, Mihala G, Rickard CM. Devices and dressings to secure peripheral venous catheters: A Cochrane systematic review and meta-analysis. Int J Nurs Stud. 2017 Feb;67:12-19. doi: 10.1016/j.ijnurstu.2016.11.007. Epub 2016 Nov 16. PMID 27889585
- [Background] Nobre A., Martins M. Prevalência de flebite da venopunção periférica: fatores associados. Revista de Enfermagem Referência 4(16): 127-138, 2018.
- [Background] Braga L. Práticas de enfermagem e a segurança do doente no processo de punção de vasos e na administração da terapêutica endovenosa (Doctoral Thesis). Universidade de Lisboa, 2017.
- [Background] Costa P. Gestão de Material Clínico de Bolso por Enfermeiros: fatores determinantes e diversidade microbiológica (Masters' Dissertation). Escola Superior de Enfermagem de Coimbra, 2017.